CLINICAL TRIAL: NCT02664519
Title: Mechanisms of Muscle Blood Flow Dysregulation and Exercise Intolerance in Chronic Kidney Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding support and not adequate number of subjects are recruited for the study
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STU 092015-005
Record Dates: First submitted 2016-01-08; First posted 2016-01-27 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Functional sympatholysis; Exercise training; Exercise intolerance; Handgrip exercise; Near infrared spectroscopy; Lower body negative pressure
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise training followed by no exercise training (Experimental): CKD subjects will be randomized to exercise training (to squeeze a tennis ball repeatedly for at least 30 min/day) or no exercise training for 28 days. Procedures in baseline visit will be repeated followed by cross over to alternate group for 28 days followed by repeat of baseline procedures.
  Interventions: Behavioral: Forearm exercise training
- No exercise training followed by exercise training (Experimental): CKD subjects will be randomized to exercise training (to squeeze a tennis ball repeatedly for at least 30 min/day) or no exercise training for 28 days. Procedures in baseline visit will be repeated followed by cross over to alternate group for 28 days followed by repeat of baseline procedures.
  Interventions: Behavioral: Forearm exercise training
- Normal Control (No Intervention): Control subjects without CKD will undergo baseline assessment as above.

INTERVENTIONS:
Behavioral: Forearm exercise training — Subjects will be asked to squeeze a tennis ball repeatedly for at least 30 min/day for 28 days at an approximate rate of 20 squeezes/min.
  Arms: Exercise training followed by no exercise training; No exercise training followed by exercise training

SUMMARY:
Patients with chronic kidney disease (CKD) experience fatigue and exercise intolerance. Increased oxidative stress in CKD may be a contributing factor. The role of impaired muscle blood flow regulation has not been fully explored. The investigators hypothesize that functional sympatholysis is exaggerated in CKD and this is associated with increased oxidative stress. The investigators also hypothesize that exercise training will improve functional sympatholysis and oxidative stress

DETAILED DESCRIPTION:
Progressive muscle weakness and premature fatigue are characterize the condition of chronic kidney disease (CKD) which can be very debilitating. Mechanisms underlying exercise intolerance in CKD is not completely understood. Previous studies have demonstrated impaired skeletal muscle vasodilation during exercise in CKD patients, which may contribute to exercise intolerance. Normally, there is blunting of sympathetic mediated vasoconstriction in exercising muscle to allow for steady blood supply to exercising muscles. This phenomenon is called functional sympatholysis. Functional sympatholysis is impaired by increases in reactive oxygen specie and may be impaired in CKD.

Experiments will be performed on 2 groups of subjects 1) Normal kidney function (eGFR>90) 2) Stage 2-3 CKD (eGFR 30-89). VAsoactive medications will be held for 72 hours before study. All participants will attend a baseline study visit, which will include a physical examination, a medical history review, vital sign measurements, and blood collection. Muscle nerve activity and muscle oxygenation will be measured while the subjects perform hand grip exercise at 30% maximum voluntary contraction with and without lower body negative pressure (- 20 mmHg). Muscle blood flow will be measured before and after hand grip exercises. CKD subjects will then be randomized to exercise training (to squeeze a tennis ball repeatedly for at least 30 min/day) or no exercise training for 28 days. Procedures in baseline visit will be repeated followed by cross over to alternate group for 28 days followed by repeat of baseline procedures. Blood flow, muscle oxygenation and muscle nerve activity will be compared between CKD and normal subjects as well as before and after exercise training for CKD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive adults
* CKD 2-3

Exclusion Criteria:

* Blood Pressure ≥140/90
* eGFR >60ml/min/1.73 m2 or eGFR <30ml/min/1.73 m2
* Any evidence of cardiopulmonary disease, left ventricular hypertrophy or systolic dysfunction by echocardiography.
* Diabetes mellitus or other systemic illness
* Pregnancy
* Any history of substance abuse or current cigarette use
* Any history of psychiatric illness
* History of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Change in muscle oxygenation | After 28 days
  Tissue oxygenation will be recorded using Near-infrared spectroscopy (NIRS)

SECONDARY OUTCOMES:
Change in Forearm vascular conductance (FVC) | After 28 days
  Doppler ultrasonography to measure blood flow
Change in plasma isoprostanes | After 28 days
  Plasma isoprostanes will be used as a measure of oxidative stress
Change in muscle sympathetic nerve activity (MSNA) | After 28 days
  MSNA will be measured using tiny tungsten wire inserted into the common peroneal nerve below fibular head.

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Result] Moore GE, Painter PL, Brinker KR, Stray-Gundersen J, Mitchell JH. Cardiovascular response to submaximal stationary cycling during hemodialysis. Am J Kidney Dis. 1998 Apr;31(4):631-7. doi: 10.1053/ajkd.1998.v31.pm9531179.
- [Result] Adams GR, Vaziri ND. Skeletal muscle dysfunction in chronic renal failure: effects of exercise. Am J Physiol Renal Physiol. 2006 Apr;290(4):F753-61. doi: 10.1152/ajprenal.00296.2005. PMID 16527920
- [Result] Paglialonga F, Lopopolo A, Scarfia RV, Galli MA, Consolo S, Brivio A, Grassi MR, Salera S, Edefonti A. Correlates of exercise capacity in pediatric patients on chronic hemodialysis. J Ren Nutr. 2013 Sep;23(5):380-6. doi: 10.1053/j.jrn.2013.04.006. Epub 2013 Jun 22. PMID 23800461
- [Result] Bradley JR, Anderson JR, Evans DB, Cowley AJ. Impaired nutritive skeletal muscle blood flow in patients with chronic renal failure. Clin Sci (Lond). 1990 Sep;79(3):239-45. doi: 10.1042/cs0790239. PMID 2169372
- [Result] Sakkas GK, Ball D, Mercer TH, Sargeant AJ, Tolfrey K, Naish PF. Atrophy of non-locomotor muscle in patients with end-stage renal failure. Nephrol Dial Transplant. 2003 Oct;18(10):2074-81. doi: 10.1093/ndt/gfg325. PMID 13679483
- [Result] Hansen J, Sander M, Thomas GD. Metabolic modulation of sympathetic vasoconstriction in exercising skeletal muscle. Acta Physiol Scand. 2000 Apr;168(4):489-503. doi: 10.1046/j.1365-201x.2000.00701.x. PMID 10759586
- [Result] Vongpatanasin W, Wang Z, Arbique D, Arbique G, Adams-Huet B, Mitchell JH, Victor RG, Thomas GD. Functional sympatholysis is impaired in hypertensive humans. J Physiol. 2011 Mar 1;589(Pt 5):1209-20. doi: 10.1113/jphysiol.2010.203026. Epub 2011 Jan 4. PMID 21224235
- [Result] Mizuno M, Iwamoto GA, Vongpatanasin W, Mitchell JH, Smith SA. Exercise training improves functional sympatholysis in spontaneously hypertensive rats through a nitric oxide-dependent mechanism. Am J Physiol Heart Circ Physiol. 2014 Jul 15;307(2):H242-51. doi: 10.1152/ajpheart.00103.2014. Epub 2014 May 9. PMID 24816260
- [Result] Piantadosi CA, Hemstreet TM, Jobsis-Vandervliet FF. Near-infrared spectrophotometric monitoring of oxygen distribution to intact brain and skeletal muscle tissues. Crit Care Med. 1986 Aug;14(8):698-706. doi: 10.1097/00003246-198608000-00007. PMID 3013501
- [Result] Kumar S, Seward J, Wilcox A, Torella F. Influence of muscle training on resting blood flow and forearm vessel diameter in patients with chronic renal failure. Br J Surg. 2010 Jun;97(6):835-8. doi: 10.1002/bjs.7004. PMID 20309951